CLINICAL TRIAL: NCT00415064
Title: An Open-Label Phase I Study of the Safety of Perifosine in Combination With Lenalidomide and Dexamethasone for Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Phase I Study of Perifosine + Lenalidomide and Dexamethasone for Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AEterna Zentaris (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Perifosine 127
Record Dates: First submitted 2006-12-20; First posted 2006-12-22 (Estimated); Last update posted 2012-07-06 (Estimated); Status verified 2011-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Perifosine; Lenalidomide; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma | interventions — perifosine; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Perifosine — Perifosine given in either 50 mg or 100 mg / day
Drug: Lenalidomide — Lenalidomide given in either 15 or 25 mg / day
Drug: Dexamethasone — Dexamethasone given in 20 mg / day

SUMMARY:
This is a phase I study of perifosine in combination with lenalidomide and dexamethasone for patients with relapsed or refractory multiple myeloma. The current protocol will enroll patients with relapsed or refractory multiple myeloma requiring second or third line therapy. Six patients each will be treated with at one of 4 dose levels in a phase 1 study. All patients will receive perifosine, lenalidomide and dexamethasone of each 28 day cycle. The doses of perifosine and lenalidomide will be varied in each group. The dose of dexamethasone will remain constant.

DETAILED DESCRIPTION:
This is a phase I study of perifosine in combination with lenalidomide and dexamethasone for patients with relapsed or refractory multiple myeloma. All patients will receive lenalidomide daily for days 1 to 21 of each 28 day cycle. Perifosine will be given daily qhs with food. Dexamethasone will be given on days 1-4, 9-12 and 17-20 for 4 cycles. After 4 cycles dexamethasone will be given only on days 1-4. Four dose levels will be studied:

1. Perifosine 50 mg, lenalidomide 15 mg and dexamethasone 20 mg
2. Perifosine 50 mg, lenalidomide 25 mg and dexamethasone 20 mg
3. Perifosine 100 mg, lenalidomide 15 mg and dexamethasone 20 mg
4. Perifosine 100 mg, lenalidomide 25 mg and dexamethasone 20 mg

Six patients will be enrolled at each dose level until the maximum tolerated dose (MTD) is reached. Six additional patients will be treated at the MTD.

ELIGIBILITY:
Inclusion Criteria:

* Subject was previously diagnosed with multiple myeloma based on standard diagnostic criteria, as follows.
* Major criteria:

  1. Plasmacytomas on tissue biopsy.
  2. Bone marrow plasmacytosis (> 30% plasma cells).
  3. Monoclonal immunoglobulin spike on serum electrophoresis immunoglobulin G (IgG) >3.5 g/dL or immunoglobulin A (IgA) > 2.0 g/dL; kappa or lambda light chain excretion > 1 g/day on 24 hour urine protein electrophoresis.
* Patients must have relapsed or refractory disease (refractory is defined as progression during treatment or within 60 days after the completion of treatment) requiring 2nd or 3rd line therapy
* Patients refractory to a combination of lenalidomide and dexamethasone will not be eligible. Patients may have received lenalidomide and/or dexamethasone

Exclusion Criteria:

* Renal insufficiency (serum creatinine levels > 3 mg/dL)..
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to perifosine (miltefosine or edelfosine).
* Known hypersensitivity to thalidomide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Every cycle

SECONDARY OUTCOMES:
Clinically significant changes in the patient's physical examination, vital signs, and clinical laboratory results | Every 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej J Jakubowiak, MD, PhD, Study Chair — University of Michigan
Locations (1):
- Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Jakubowiak AJ, Richardson PG, Zimmerman T, Alsina M, Kaufman JL, Kandarpa M, Kraftson S, Ross CW, Harvey C, Hideshima T, Sportelli P, Poradosu E, Gardner L, Giusti K, Anderson KC. Perifosine plus lenalidomide and dexamethasone in relapsed and relapsed/refractory multiple myeloma: a Phase I Multiple Myeloma Research Consortium study. Br J Haematol. 2012 Aug;158(4):472-80. doi: 10.1111/j.1365-2141.2012.09173.x. Epub 2012 May 29. PMID 22640031